CLINICAL TRIAL: NCT04046328
Title: A Phase IIa, Proof of Concept, Randomized, Double-Blind, Dose-Finding, Cross-Over Study of the Efficacy, Safety and Tolerability of a New Enteric-Coated Cholestyramine Capsule in Adult Short Bowel Syndrome Patients
Brief Title: Efficacy, Safety and Tolerability of Enteric-Coated Cholestyramine Capsules for Adult Short Bowel Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult recruitment
Sponsor: Pharmascience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMS-2018-002; 2018-004419-32 (EudraCT Number)
Record Dates: First submitted 2019-07-26; First posted 2019-08-06 (Actual); Results first posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — Capsules

STUDY DESIGN:
Intervention Model Description: Multiple-center, randomized, double-blind, double dummy, 2-period, 2-sequence cross-over design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be fully blinded, using the double dummy technique (combination of active ECC capsules and matching placebo in the low dose treatment arm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- "Low" Dose ECC Regimen (Experimental): ECC at the 1.7 g daily dose, administered BID (twice daily) as 2 capsules of ECC, plus 3 capsules of placebo, at least 30 minutes before breakfast and 2 capsules of ECC, plus 3 capsules of placebo at least 30 minutes before evening meal.
  Interventions: Drug: Enteric-Coated Cholestyramine (ECC) Capsule; Drug: Placebo
- "High" Dose ECC Regimen (Experimental): ECC at the 4.25 g daily dose, administered BID (twice daily) as 5 capsules of ECC at least 30 minutes before breakfast and 5 capsules of ECC at least 30 minutes before evening meal.
  Interventions: Drug: Enteric-Coated Cholestyramine (ECC) Capsule

INTERVENTIONS:
Drug: Enteric-Coated Cholestyramine (ECC) Capsule — Enteric-Coated Delayed Release Cholestyramine Capsules
Drug: Placebo — Enteric-Coated Delayed Release Placebo Capsules
  Arms: "Low" Dose ECC Regimen

SUMMARY:
A new Enteric-Coated Cholestyramine (ECC) capsule has been developed to manage diarrhea associated with Short Bowel Syndrome (SBS) in adults. The formulation is expected to release cholestyramine in the remaining segment of the small intestine in SBS patients, thus binding bile acids after fat digestion, but before induction of diarrhea in the colon. The delayed-release profile is also expected to help reduce the potential for drug-drug interactions occurring in the proximal small intestine. Two doses of ECC will be studied for efficacy, safety and tolerability in this Phase IIa trial.

DETAILED DESCRIPTION:
A new Enteric-Coated Cholestyramine (ECC) capsule has been developed to manage diarrhea associated with Short Bowel Syndrome (SBS). SBS is usually caused by the significant resection or loss of function of the ileum, leading to reduced reabsorption of bile acids and subsequent osmotic diarrhea. The new ECC formulation could release cholestyramine in the remaining segment of the small intestine in SBS patients, delivering and binding bile acids before they induce diarrhea in the colon. The proposed advantages of this formulation are: a) to prevent drug-drug interactions in the proximal GI tract, b) to preserve the fat digestive properties of bile acids in the duodenum and 3) to offer a more palatable dosage form to patients. Moreover, since distal delivery of cholestyramine is expected to be more effective in diarrhea prevention/reduction in SBS, lower doses than the ones used with non-enteric coated cholestyramine may be sufficient. Two doses of ECC will be studied for efficacy, safety and tolerability in well-defined non fully-colectomized, adult SBS patients suffering from diarrhea.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, ambulatory male and female subjects
2. Provision of signed and dated informed consent form (ICF)
3. Age ≥ 18 years and ≤ 80 years
4. Stable SBS of:

   1. Non-surgical origin; OR
   2. Surgical origin where the last surgical ileal resection was performed at least 6 months prior to enrolment
5. Partial, Home Parenteral Nutrition and/or parenteral fluids are allowed, at a maximum frequency of 6 times a week throughout the trial, as long as the regimen has been stable for at least 2 weeks prior to screening and is expected to remain unchanged during the study
6. At least 50 % of the colon being intact
7. Intact duodenum
8. BMI ≥ 18
9. Presence of stable chronic diarrhea for at least 3 months prior to enrolment as evidenced by medical history
10. Presence of stable chronic diarrhea during the 2-week screening diary period before randomization, as evidenced by completion of a screening diary demonstrating:

    1. Mean daily production of at least 3 soft or watery stools (BSFS scores 6 or 7); or
    2. More than 3 bowel movements per day on average with >25% of them being BSFS type 6 or 7
11. Stated willingness and ability to comply with all study procedures, including daily recording of bowel movements and BSFS in the patient diaries, and availability for the duration of the study
12. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without clinical significance, as determined by the investigator
13. Female subjects must meet one of the following criteria:

    a) Participant is of childbearing potential and agrees to use one of the accepted contraceptive regimens from at least 30 days prior to the first study treatment administration through to at least 30 days after the last dose of the study treatment. An acceptable method of contraception includes one of the following:
    1. Abstinence from heterosexual intercourse
    2. Systemic contraceptives (combined birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
    3. Intrauterine device (with or without hormones)
    4. Condom with spermicide

    b) Participants of non-childbearing potential, defined as surgically sterile (i.e. has undergone complete hysterectomy or bilateral oophorectomy) or is in a menopausal state (i.e. at least 1 year without menses prior to the first study drug administration) are eligible

Exclusion Criteria:

1. Patients with known or suspected intestinal strictures of clinical relevance as judged by the Investigator
2. Active inflammatory bowel disease (IBD) or fistula during the screening period as judged by the Investigator
3. Crohn's disease patients not being in clinical remission for the last 12 weeks prior to randomization
4. Diarrhea caused by other causes than SBS
5. Presence of clinically significant steatorrhea, requiring pancreatic enzymes supplementation
6. Presence of complete biliary obstruction
7. Presence of active cancer (except resected cutaneous basal or squamous cell carcinoma and except in situ cervical cancer) and/or need to receive chemotherapy or radiotherapy during the study
8. History of allergic reaction to cholestyramine or any excipient of the investigational drug product or placebo, or packaging components
9. Females who are lactating at screening
10. Females who are pregnant according to the pregnancy test at screening or prior to the first study treatment administration
11. Significant history (at least 3 consecutive months in the year prior to Screening) of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
12. Subjects who took an Investigational Product (IP) in the 30 days prior to the first study drug administration
13. Any other clinically significant condition that is considered by the principal investigator as being susceptible to put the patient at greater safety risk, influence response to study product, or interfere with study assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marek Kunecki, MD, PhD, Principal Investigator — Wojewódzki Specjalistyczny Szpital im. M. Pirogowa w Łodzi; Konrad Matysiak, MD, PhD, Principal Investigator — Solumed Centrum Medyczne; Kinga Szczepanek, MD, Principal Investigator — Szpital Wielospecjalistyczny im. Stanleya Dudricka
Locations (3):
- Poland (3):
  - Wojewódzki Specjalistyczny Szpital im. M. Pirogowa w Łodzi, Lodz
  - Solumed Centrum Medyczne, Poznan
  - Szpital Wielospecjalistyczny im. Stanleya Dudricka, Skawina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a multiple center, randomized, double-blind, double dummy, 2-period, 2-sequence cross-over study design planned to evaluate 18 patients at three study centers. Due to early study termination only 13 patients were randomized and received treatment with ECC.
Groups:
- "Low" Dose ECC Regimen, Then "High" Dose ECC Regimen: "Low" Dose: ECC at the 1.7 g daily dose, administered BID as 2 capsules of ECC, plus 3 capsules of placebo, at least 30 minutes before breakfast and 2 capsules of ECC, plus 3 capsules of placebo at least 30 minutes before evening meal.
  "High" Dose: ECC at the 4.25 g daily dose, administered BID as 5 capsules of ECC at least 30 minutes before breakfast and 5 capsules of ECC at least 30 minutes before evening meal.
  Enteric-Coated Cholestyramine (ECC) Capsule: Enteric-Coated Delayed Release Cholestyramine Capsules
  Placebo: Enteric-Coated Delayed Release Placebo Capsules
- "High" Dose ECC Regimen, Then "Low" Dose ECC Regimen: "High" Dose: ECC at the 4.25 g daily dose, administered BID as 5 capsules of ECC at least 30 minutes before breakfast and 5 capsules of ECC at least 30 minutes before evening meal.
  "Low" Dose: ECC at the 1.7 g daily dose, administered BID as 2 capsules of ECC, plus 3 capsules of placebo, at least 30 minutes before breakfast and 2 capsules of ECC, plus 3 capsules of placebo at least 30 minutes before evening meal.
  Enteric-Coated Cholestyramine (ECC) Capsule: Enteric-Coated Delayed Release Cholestyramine Capsules
  Placebo: Enteric-Coated Delayed Release Placebo Capsules
Period: First Intervention (14 Days)
Arm/Group | "Low" Dose ECC Regimen, Then "High" Dose ECC Regimen | "High" Dose ECC Regimen, Then "Low" Dose ECC Regimen
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | "Low" Dose ECC Regimen, Then "High" Dose ECC Regimen | "High" Dose ECC Regimen, Then "Low" Dose ECC Regimen
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0
Period: Second Intervention (14 Days)
Arm/Group | "Low" Dose ECC Regimen, Then "High" Dose ECC Regimen | "High" Dose ECC Regimen, Then "Low" Dose ECC Regimen
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intent-to-Treat (ITT Population): Demographics and baseline characteristics were assessed for the overall ITT Population
Arm/Group | Intent-to-Treat (ITT Population)
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (15.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0
  Black | 0
  Caucasian | 13
  Other | 0
Region of Enrollment [Number; unit: participants]
  Poland | 13
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.1 (3.84)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Weekly Frequency of Bowel Movements Measured Between Baseline and the Second Week of Treatment
Description: Change in the weekly frequency of bowel movements measured between baseline and the second week of treatment. Baseline is defined as the second week of screening for treatment period 1 and second week of washout for treatment period 2.
Time Frame: Baseline and Week 2 of treatment (Days 8 to 14, and Days 36 to 42)
Measure: Mean (Standard Deviation); unit: Weekly bowel movements
Groups:
- "Low" Dose ECC Regimen: ECC at the 1.7 g daily dose, administered BID as 2 capsules of ECC, plus 3 capsules of placebo, at least 30 minutes before breakfast and 2 capsules of ECC, plus 3 capsules of placebo at least 30 minutes before evening meal.
  Enteric-Coated Cholestyramine (ECC) Capsule: Enteric-Coated Delayed Release Cholestyramine Capsules
  Placebo: Enteric-Coated Delayed Release Placebo Capsules
- "High" Dose ECC Regimen: ECC at the 4.25 g daily dose, administered BID as 5 capsules of ECC at least 30 minutes before breakfast and 5 capsules of ECC at least 30 minutes before evening meal.
  Enteric-Coated Cholestyramine (ECC) Capsule: Enteric-Coated Delayed Release Cholestyramine Capsules
Arm/Group | "Low" Dose ECC Regimen | "High" Dose ECC Regimen
Number analyzed (Participants) | 13 | 13
Weekly bowel movements | -11.5 (11.38) | -13.4 (9.73)

2. Secondary Outcome: Total Number of Bowel Movements for the Whole 2-week Treatment Period
Time Frame: Days 1 to 14 and Days 29 to 42
Measure: Mean (Standard Deviation); unit: Bowel movements
Arm/Group | "Low" Dose ECC Regimen | "High" Dose ECC Regimen
Number analyzed (Participants) | 13 | 13
Bowel movements | 52.5 (20.12) | 55.1 (25.18)

3. Secondary Outcome: Mean Daily Stool Form Score According to the BSFS (Bristol Stool Form Scale), Measured During the Second Week of Treatment
Description: The BSFS classifies the form of human feces into seven categories (Type 1 to Type 7) based on stool shape and consistency. Types or scores of 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, 5 tending towards diarrhea, and 6 and 7 indicate diarrhea.
Time Frame: Days 8 to 14, and Days 36 to 42
Measure: Mean (Standard Deviation); unit: Score on BSFS scale
Arm/Group | "Low" Dose ECC Regimen | "High" Dose ECC Regimen
Number analyzed (Participants) | 13 | 13
Score on BSFS scale | 3.6 (1.42) | 3.7 (1.76)

4. Secondary Outcome: Mean Daily Dose of Loperamide in mg, if Used, During the Second Week of Treatment
Time Frame: Days 8 to 14, and Days 36 to 42
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | "Low" Dose ECC Regimen | "High" Dose ECC Regimen
Number analyzed (Participants) | 7 | 7
mg | 72.9 (43.05) | 68.9 (53.19)

ADVERSE EVENTS:
Time Frame: From patient randomization to the end of study visit, approximately 44 days
Arm/Group | "Low" Dose ECC Regimen | "High" Dose ECC Regimen
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 3/13 | 4/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | "Low" Dose ECC Regimen (N=13) | "High" Dose ECC Regimen (N=13)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 1
Pulpitis dental (Infections and infestations) | 1 | 1
C-reactive protein increased (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed and abbreviated statistical analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the study results by the Investigator, the Center and by any member of the Investigational Team shall require a prior express approval of Pharmascience in writing.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT04046328/Prot_SAP_000.pdf